CLINICAL TRIAL: NCT02895997
Title: Turning Night Into Day: Transcontinental Provision of Telehealth By and For the Emory Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Timothy G. Buchman, PhD, MD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00088367
Record Dates: First submitted 2016-09-01; First posted 2016-09-12 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Mental Fatigue
Keywords: mental fatigue; critical care
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Operations Room Staff (Experimental): Clinicians and critical care nurse volunteers from the clinical operations room (COR) staff at Emory University Hospital will travel to Sydney Australia to deliver telemedicine.
  Interventions: Other: Travel Telehealth Delivery

INTERVENTIONS:
Other: Travel Telehealth Delivery — Clinical Operations Room (COR) staff will travel to Sydney Australia to deliver telehealth to patients in Georgia United States. Upon arrival, participants will have eight nights and seven days free of clinical responsibilities. Thereafter, each participant will work four consecutive days of 12 hour shifts followed by four consecutive days with no clinical assignment. The following week, participants will work three consecutive days of 12 hour shifts followed by four consecutive days with no clinical assignment. Upon return to the USA, participants will have a week free of clinical responsibilities.

SUMMARY:
The purpose of the study is to determine if temporarily relocating clinicians who deliver remote care using the eICU telehealth system to Sydney, Australia will lead to greater job satisfaction, reduced physiologic stress, and improve performance. Four nurses and six physicians will be sent to a site in Sydney Australia on a rotating basis to determine whether providing care during the Australian daytime is more efficient and precise than providing care during the night in the United States.

DETAILED DESCRIPTION:
The purpose of the study is to determine if temporarily relocating clinicians who deliver remote care using the eICU telehealth system to Sydney Australia will lead to greater job satisfaction, reduced physiologic stress, and improve performance. Four nurses and six physicians will be sent to a site in Sydney Australia on a rotating basis to determine whether providing care during the Australian daytime is more efficient and precise than providing care during the night in the United States.

As part of this pilot, each participant will undergo a series of evaluations before leaving, while in Australia, and after returning. The evaluations will include questionnaires related to well-being, task assessment (such as completing a paper maze or performing arithmetic), physiology assessment (such as continuous measure of heart rate by a wristwatch type device), and stress assessment (by sampling saliva and measuring cortisol and interleukin-1 Beta).

The researchers would like to determine whether normalization of the provider's (physician or nurse who are the research subjects) sleep-wake cycle improves subjective and objective well-being. Additionally, investigators seek to determine whether normalization of the provider's (physician or nurse who are the research subjects) sleep-wake cycle improves alertness and focus, and determine whether normalization of the provider's (physician or nurse who are the research subjects) sleep-wake cycle improves job performance.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians working in the clinical operations room at Emory University Hospital who volunteer participation in the study

Exclusion Criteria:

* Declining to participate after the first phase of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Cortisol Levels | Baseline, Post Intervention (Up to 8 weeks)
  Saliva will be collected via a mouth swab and tested for cortisol levels. Cortisol is a stress biomarker.

SECONDARY OUTCOMES:
Change in Stanford Sleepiness Scale Score | Baseline, Post Intervention (Up to 8 weeks)
  The Stanford Sleepiness Scale is a seven point scale that asks participants to assess how alert they are feeling throughout the day. A result of 4 or below may indicate that a participant could be suffering from a lack of sleep
Change in the Trail Making Test A Score | Baseline, Post Intervention (Up to 8 weeks)
  During the Trail Making Test A, participants will be asked to draw lines to connect circled numbers in a numerical sequence (i.e., 1-2-3, etc.) as rapidly in possible. A shorter time indicates better cognition.
Change in the Trail Making Test B Score | Baseline, Post Intervention (Up to 8 weeks)
  During the Trail Making Test B, participants will be asked to draw lines to connect circled numbers and letters in an alternating numeric and alphabetic sequence (i.e., 1-A-2-B, etc.) as rapidly as possible. A shorter time indicates better cognition.
Change in Physical Activity assessed by Multi-Scale Entropy | Baseline, Post Intervention (Up to 8 weeks)
  Multi-scale entropy will be measured using a Jawbone wristband device provided to participants upon enrollment.
Change in Physical Activity assessed by Multi-Scale Complexity | Baseline, Post Intervention (Up to 8 weeks)
  Multi-scale complexity will be measured using a Jawbone wristband device provided to participants upon enrollment.
Change in Heart Rate Variability assessed by Deceleration Capacity | Baseline, Post Intervention (Up to 8 weeks)
  Deceleration capacity will be measured using a Jawbone wristband device provided to participants upon enrollment.
Change in Heart Rate Variability assessed by Acceleration Capacity | Baseline, Post Intervention (Up to 8 weeks)
  Acceleration capacity will be measured using a Jawbone wristband device provided to participants upon enrollment.
Frequency of Arrhythmias | Duration of Study (Up to 31 Days)
  The frequency of arrhythmias will be collected using a Jawbone wristband device provided to participants upon enrollment.
Change in Sleep Latency | Baseline, Post Intervention (Up to 8 weeks)
  Sleep latency is the length of time it takes to accomplish the transition from full wakefulness to sleep. This will be measured in minutes using a Jawbone wristband device provided to participants upon enrollment.
Number of Awakenings per Hour | Duration of Study (Up to 31 Days)
  The number of times a participants awakes during sleep will be monitored at every hour using a Jawbone wristband device provided to participants upon enrollment.
Change in Percent of Non Rapid Eye Movement (REM) Sleep | Baseline, Post Intervention (Up to 8 weeks)
  Change is the difference between the percentage of non REM sleep taken during performance phases.
Change in Mood Symptom Questionnaire Score | Baseline, Post Intervention (Up to 8 weeks)
  The Mood Symptom Questionnaire was originally designed to diagnose bipolar disorder. The questionnaire takes about five minutes to complete, and can provide important insights into diagnosis and treatment.If the patient answers "Yes" to seven or more of the 13 items in question number 1 AND "Yes" to question number 2 AND "Moderate" or "Serious" to question number 3, there is a positive screen.
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline, Post Intervention (Up to 8 weeks)
  The PHQ-9 is a multi-purpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. A score of 5-9 represents signs of minimal depression symptoms. A score of 10-14 represents symptoms of minor depression. A score of 15-19 represents symptoms of major depression, moderately severe. A score of greater than 20 represents symptoms of major depression, severe.
Change in Number of Camera Sessions | Day 1, Day 31
  Difference in the number of camera sessions completed during performance phases.
Change in Duration of Camera Sessions | Day 1, Day 31
  Difference in the duration of camera sessions during performance phases measured in minutes.
Change in Urgency of Clinical Contacts | Day 1, Day 31
  Difference in priority levels assigned to each clinical contact (levels: preventative; informative/procedural; urgent; life-threatening)
Change in Number if Clinical Record Entries | Day 1, Day 31
  Difference in the number of clinical record entries made by physicians only during the performance phases.
Change in Duration of Service | Day 1, Day 31
  Difference in the duration of physician services during each performance phase measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Buchman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with future researchers.